CLINICAL TRIAL: NCT04618380
Title: Premium Monovision Versus Bilateral Myopic Monovision, Hybrid Monovision and Bilateral Trifocal Implantation. A Comparative Study.
Brief Title: Premium Monovision Versus Other Types of Monovision and Bilateral Trifocal Implantation.
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES13/Th9/22-10-2020
Record Dates: First submitted 2020-11-01; First posted 2020-11-05 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Presbyopia; Refractive Errors; Cataract
Keywords: pseudophakic presbyopic correction; premium monovision; myopic monovision; multifocal intraocular lenses; hybrid monovision
MeSH Terms: conditions — Presbyopia; Refractive Errors; Cataract | interventions — Contrast Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bilateral trifocal implantation: Bilateral implantation of trifocal diffractive intraocular lenses (Panoptix, Alcon) targeting emmetropia
  Interventions: Diagnostic Test: bUD-VA,bUN-RA, bUI-RA, bUI-CPS, bUN-CPS, contrast sensitivity
- Myopic monovision: The dominant eye defocus is targeted to -0.50 diopters while the recessive one to -1.25 diopters with bilateral implantation of monofocal intraocular lenses (SN60WF, Alcon)
  Interventions: Diagnostic Test: bUD-VA,bUN-RA, bUI-RA, bUI-CPS, bUN-CPS, contrast sensitivity
- Hybrid monovision: Hybrid monovision combines a monofocal intraocular (SN60WF, Alcon) in the dominant eye and a trifocal diffractive intraocular lens (Panoptix, Alcon) in the recessive one
  Interventions: Diagnostic Test: bUD-VA,bUN-RA, bUI-RA, bUI-CPS, bUN-CPS, contrast sensitivity
- Premium monovision: Participants received a bifocal hybrid (refractive at the centre, diffractive at the periphery) intraocular lens (Restor +2.50 diopters, Alcon) in the dominant eye and a trifocal diffractive intraocular lens (Panoptix, Alcon) in the recessive one, targeting emmetropia in both eyes.
  Interventions: Diagnostic Test: bUD-VA,bUN-RA, bUI-RA, bUI-CPS, bUN-CPS, contrast sensitivity

INTERVENTIONS:
Diagnostic Test: bUD-VA,bUN-RA, bUI-RA, bUI-CPS, bUN-CPS, contrast sensitivity — The following clinical indexes are evaluated:
  1. Binocular uncorrected distant visual acuity (bUD-VA) using the Greek version of the Early Treatment Diabetic Retinopathy Study Chart at four meters distance
  2. Binocular uncorrected reading acuity at 60cm (bUI-RA) and at 40cm (bUN-RA), and
  3. Binocular uncorrected critical print size at 60cm (bUI-CPS) and at 40cm (bUN-CPS).
  All near and intermediate vision parameters are obtained using the Democritus Digital Acuity Reading Test (DDART), which is based on the Greek version of MNREAD.
  Contrast sensitivity are evaluated with the Pelli-Robson test.

SUMMARY:
Primary objective of this study was to compare the efficacy of premium monovision with Restor and Panoptix, against other prevalent monovision techniques and against bilateral Panoptix implantation in a sample of patients following lens-extraction surgery.

DETAILED DESCRIPTION:
Four study groups were formed according to the procedure and the intraocular lens technology that was used: a) Monovision Group (MoG), b) Multifocal Lens Group (MfG), c) Hybrid Monovision Group (HmG), and, d) Premium Monovision Group (PmG). Patients who have undergone one of the above categories of presbyopia correction surgery were selected to compare the effectiveness of these techniques by evaluating the uncorrected near, intermediate and distant visual acuity as well as the degree of subjective patient satisfaction, contrast sensitivity, dysphotopsia symptoms and spectacle independence .

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of senile cataract with stage 2 nuclear opalescence according to the Lens Opacities Classification System III (LOCS-3) grading scale

Exclusion Criteria:

* Manifest astigmatism > 1.00 diopters
* Reports of headaches and/or eyestrain associated with visual activities
* Positive, pathologic ocular cover test (near & distant) and / or the Mallett's disparity test (near & distant) and the double Maddox rod test
* Endothelial cell count less than 1900/mm2
* Glaucoma
* intraocular pressure-lowering medications
* Former incisional surgery
* Former diagnosis of corneal disease
* Former diagnosis of fundus disease
* Diabetes
* Autoimmune diseases
* Mental diseases

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from the Cataract Service of the University Hospital of Alexandroupolis in a consecutive-if-eligible basis.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Binocular uncorrected distant visual acuity [bUD-VA] | through study completion, an average of 2.5years
  bUD-VA is obtained using the Greek version of the Early Treatment Diabetic Retinopathy Study Chart at four meters distance. This parameter is obtained six months following the operation of the second eye.
Binocular uncorrected intermediate reading acuity (at 60cm) [bUI-RA)] | through study completion, an average of 2.5years
  bUI-RA is obtained using the DDART reading test, which is based on the Greek version of MNREAD. This parameter is obtained six months following the operation of the second eye.
binocular uncorrected near reading acuity (at 40cm) [bUN-RA] | through study completion, an average of 2.5years
  bUN-RA is obtained using the DDART reading test, which is based on the Greek version of MNREAD. This parameter is obtained six months following the operation of the second eye.
binocular uncorrected intermediate critical print size (at 60cm) [bUI-CPS] | through study completion, an average of 2.5years
  bUI-CPS is obtained using the DDART reading test, which is based on the Greek version of MNREAD. This parameter is obtained six months following the operation of the second eye.
binocular uncorrected near critical print size (at 40cm )[bUN-CPS] | through study completion, an average of 2.5years
  bUN-CPS is obtained using the DDART reading test, which is based on the Greek version of MNREAD. This parameter is obtained six months following the operation of the second eye.

SECONDARY OUTCOMES:
Dysphotopsia symptoms | through study completion, an average of 2.5years
  Dysphotopsia is evaluated with two direct 4-scale, Likert-type questions (Always, Most of the times, Sometimes, Never) pertaining on the subjective perception of glare and unwanted shadows. This parameter is obtained six months following the operation of the second eye.
Contrast sensitivity | through study completion, an average of 2.5years
  Contrast sensitivity is evaluated with the Pelli-Robson test. This parameter is obtained six months following the operation of the second eye.
Spectacle independence | through study completion, an average of 2.5years
  Spectacle dependence is also evaluated for both distant and near vision by two direct 4-scale Likert-type questions (Always, Most of the times, Sometimes, Never). This parameter is obtained six months following the operation of the second eye.
Subjective satisfaction using Visual Function Index (VF-14 instrument) (total score, VF14-NV score & VF14-DV score) | through study completion, an average of 2.5years
  Subjective satisfaction rates are assessed using the prevalent VF-14 instrument. Further to the total VF-14 score assessment, two additional scores are calculated: a) Near vision VF score (VF14-NV) derived from items that assess the perceived difficulty in near vision activities (items 1,2,3,7,8,9 and 11), and, b) Distant vision VF score (VF14-DV) derived from items that assess the perceived difficulty of distant vision activities (items 4, 5, 6, 10, 12, 13 and 14).
  VF-14 has a final score from 0 to 100. A score of 100 indicates able to do all applicable activities. A score of 0 indicates unable to do all applicable activities because of vision.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD,PHD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Result] Labiris G, Panagiotopoulou EK, Chatzimichael E, Tzinava M, Mataftsi A, Delibasis K. Introduction of a digital near-vision reading test for normal and low vision adults: development and validation. Eye Vis (Lond). 2020 Oct 22;7:51. doi: 10.1186/s40662-020-00216-0. eCollection 2020. PMID 33102611
- [Derived] Labiris G, Panagiotopoulou EK, Perente A, Ntonti P, Delibasis K, Fotiadis I, Konstantinidis A, Dardabounis D. Premium Monovision versus Bilateral Myopic Monovision, Hybrid Monovision and Bilateral Trifocal Implantation: A Comparative Study. Clin Ophthalmol. 2022 Mar 4;16:619-629. doi: 10.2147/OPTH.S351091. eCollection 2022. PMID 35282170